CLINICAL TRIAL: NCT01729871
Title: A Randomized, Open-label, Active-controlled Multi-center Study to Assess Safety of Uninterrupted Rivaroxaban vs. Usual Care in Subjects Undergoing Catheter Ablation Therapy for Atrial Fibrillation
Brief Title: A Study Exploring Two Treatment Strategies in Patients With Atrial Fibrillation Who Undergo Catheter Ablation Therapy
Acronym: VENTURE-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100732; RIVAROXAFL3002 (Other: Janssen Scientific Affairs, LLC); 2012-001484-79 (EudraCT Number)
Record Dates: First submitted 2012-10-23; First posted 2012-11-20 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Irregular heart beat; Catheter Ablation; Rivaroxaban
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rivaroxaban (Experimental): rivaroxaban 20 mg orally, once-daily, administered preferably with the evening meal
  Interventions: Drug: rivaroxaban
- vitamin K antagonist (VKA) (Experimental): dose-adjusted vitamin K antagonist (VKA) to achieve a recommended International Normalized Ratio (INR) of 2.0 to 3.0
  Interventions: Drug: uninterrupted vitamin K antagonist (VKA)

INTERVENTIONS:
Drug: rivaroxaban — rivaroxaban 20 mg orally, once-daily, administered preferably with the evening meal
  Arms: rivaroxaban
Drug: uninterrupted vitamin K antagonist (VKA) — dose-adjusted vitamin K antagonist (VKA) to achieve a recommended International Normalized Ratio (INR) of 2.0 to 3.0
  Arms: vitamin K antagonist (VKA)

SUMMARY:
The purpose of this exploratory study is to evaluate the safety of rivaroxaban and uninterrupted vitamin K antagonist (VKA) in adult participants with non-valvular atrial fibrillation (NVAF) who undergo catheter ablation as measured by post-procedure major bleeding events.

DETAILED DESCRIPTION:
This is a randomized (participants are assigned to intervention groups by chance), open-label (both physicians and participants know the identity of the assigned treatment), active-controlled, multi-center safety study of rivaroxaban or VKA before and after a catheter ablation procedure. This study requires collaboration with medical institutions that provide access to electrophysiologists who normally perform the catheter ablation procedure. In this study, NVAF is to be defined as the presence of AF in a person who does not have a prosthetic heart valve (annuloplasty with or without prosthetic ring, commissurotomy and/or valvuloplasty are permitted) and who does not have hemodynamically significant mitral valve stenosis. Approximately 250 eligible participants, age 18 years or older, with a history of paroxysmal, persistent, or long standing persistent NVAF who are scheduled to undergo an elective catheter ablation procedure will be randomized in a 1:1 ratio to receive either rivaroxaban 20 mg orally, once-daily, administered preferably with the evening meal or VKA (adjusted to achieve a recommended International Normalized Ratio of 2.0 to 3.0).

The study will consist of a screening period, a pre-procedure period, procedure period and post-procedure period. The screening period will begin up to 2 weeks prior to randomization. Participants will be randomized at the beginning of the pre-procedure period. During this period, participants will be recommended to receive their assigned treatment for at least 4 weeks (maximum of 5 weeks) before the catheter ablation procedure. For participants with the sufficient anticoagulation, documented for the 3 weeks prior to randomization, and for participants with a transesophageal echocardiogram (TEE) or intracardiac echocardiography (ICE), the length of the pre-procedure period may be reduced down to 1-7 days and must include any transition from the previous anticoagulation therapy to randomized study drug.

After the catheter ablation procedure, participants will receive their post-procedure dose of study drug through a minimum of 30 + - 5 days. In addition to scheduled visits and telephone calls the study may also include additional phone calls and visits by the participant to the site when dose adjustment is required for usual care.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for a catheter ablation procedure for non-valvular atrial fibrillation (NVAF);
* Have a documented history of paroxysmal (lasting <1 week) or persistent (lasting >1 week and <1 year or requiring pharmacological or electrical cardioversion), or long standing persistent (>=1 year) NVAF;
* Be suitable for anticoagulant therapy and catheter ablation as per the judgment of the investigator;
* Women must be postmenopausal before entry or practicing a highly effective method of birth control when heterosexually active;
* Women of childbearing potential must have a negative serum pregnancy test at screening;
* Be willing and able to adhere to the prohibitions and restrictions specified in the study protocol;
* Have a life expectancy of at least 6 months

Exclusion Criteria:

* Has a history of a prior stroke, transient ischemic attack (TIA) or non-convulsive status epilepticus within 6 months of the screening visit;
* Has a history of a major bleeding or thromboembolic event within the 12 months immediately preceding the catheter ablation procedure;
* Has had major surgery (requiring general anesthesia), within 6 months before screening or planned surgery during the time the subject is expected to participate in the study;
* Has NVAF due to electrolyte imbalance, hyperthyroidism, or other reversible or noncardiac cause of NVAF;
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (44):
- United States (24):
  - Beverly Hills, California
  - Los Angeles, California
  - Sacramento, California
  - San Francisco, California
  - Jacksonville, Florida
  - Maywood, Illinois
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Saint Louis Park, Minnesota
  - Ridgewood, New Jersey
  - Flushing, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Seattle, Washington
  - Tacoma, Washington
- Belgium (5):
  - Aalst
  - Antwerp
  - Bruges
  - Genk
  - Hasselt
- France (5):
  - Brest
  - Montpellier
  - Pessac
  - Toulouse Cedex 9 N/A
  - Vandœuvre-lès-Nancy
- Germany (7):
  - Bad Krozingen
  - Bad Nauheim
  - Berlin
  - Dresden
  - Jena
  - Mönchengladbach
  - Neuwied
- United Kingdom (3):
  - Bournemouth
  - Cottingham
  - London

REFERENCES:
- [Derived] Cappato R, Marchlinski FE, Hohnloser SH, Naccarelli GV, Xiang J, Wilber DJ, Ma CS, Hess S, Wells DS, Juang G, Vijgen J, Hugl BJ, Balasubramaniam R, De Chillou C, Davies DW, Fields LE, Natale A; VENTURE-AF Investigators. Uninterrupted rivaroxaban vs. uninterrupted vitamin K antagonists for catheter ablation in non-valvular atrial fibrillation. Eur Heart J. 2015 Jul 21;36(28):1805-11. doi: 10.1093/eurheartj/ehv177. Epub 2015 May 14. PMID 25975659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 37 sites in 5 countries.
Pre-assignment Details: 248 participants were randomized correctly to study, with an equal number of participants randomized to both treatment arms. The intention to treat (ITT) analysis set includes all participants who were correctly randomized into study. There are 5 screen failures who were not included in ITT analysis set because they were incorrectly randomized.
Groups:
- Rivaroxaban: Participants were received Rivaroxaban 20 milligram (mg) orally once-daily administered preferably with the evening meal for 8-10 weeks.
- Vitamin K Antagonist: Participants were received dose-adjusted vitamin K antagonist (VKA) to achieve a recommended International Normalized Ratio (INR) of 2.0 to 3.0 for 8-10 weeks.
Period: Overall Study
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Started | 124 | 124
Completed | 112 | 101
Not Completed | 12 | 23
Not completed — Adverse Event | 7 | 7
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Vitamin K Antagonist | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.86) | 60.5 (10.51) | 59.5 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 86 | 90 | 176
Region of Enrollment [Number; unit: participants]
  Belgium | 24 | 24 | 48
  France | 19 | 19 | 38
  Germany | 18 | 19 | 37
  Great Britain | 24 | 24 | 48
  United States of America | 39 | 38 | 77
Race [Number; unit: participants]
  ASIAN | 5 | 2 | 7
  BLACK | 3 | 3 | 6
  N/A | 4 | 3 | 7
  WHITE | 112 | 116 | 228
Ethnicity [Number; unit: participants]
  HISPANIC/LATINO | 0 | 4 | 4
  N/A | 34 | 26 | 60
  NOT HISPANIC/LATINO | 90 | 94 | 184
Body-Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (5.74) | 28.9 (5.49) | 29.4 (5.62)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81 (9.85) | 79.4 (10.78) | 80.2 (10.34)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 133.3 (15.6) | 131.2 (17.68) | 132.2 (16.67)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Post-Procedure Major Bleeding Events
Description: Post-procedure major bleeding events include Thrombolysis in Myocardial Infarction (TIMI), International Society on Thrombosis and Haemostasis (ISTH) and Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) Severe/life threatening bleeding.
Time Frame: Up to 30 plus or minus (+-) 5 days after the catheter ablation procedure
Population: Per-protocol analysis set included all randomized participants who took at least 1 dose of study drug and had undergone the catheter ablation procedure.
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Number analyzed (Participants) | 114 | 107
Participants
  TIMI Major Bleeding | 0 | 0
  ISTH Major Bleeding | 0 | 1
  GUSTO Severe/Life Threatening Bleeding | 0 | 0

2. Secondary Outcome: Number of Participants With Composite Endpoint of Myocardial Infarction (MI), Ischemic Stroke, Non-Central Nervous System (Non-CNS) Systemic Embolism and Vascular Death
Description: The composite endpoint include Myocardial Infarction (MI), Ischemic Stroke, Non-Central Nervous System (non-CNS) Systemic Embolism and Vascular Death.
Time Frame: Up to 30 plus or minus (+-) 5 days after the catheter ablation procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Number analyzed (Participants) | 114 | 107
Participants | 0 | 2

3. Secondary Outcome: Number of Participants With Myocardial Infarction (MI)
Description: The MI was defined as clinical symptoms consistent with myocardial ischemia and cardiac biomarker elevation greater than the site's upper limit of normal (ULN) or development of new pathological Q waves in at least 2 contiguous leads on the electrocardiogram (ECG) or autopsy confirmation, OR Creatine kinase-muscle and brain subunit [or creatine kinase (CK) in the absence of CK-MB] greater than (>) 3 or 5 or 10 x ULN for samples obtained within 24 hours of the procedure if the baseline values were normal or at least a 50 percent (%) increase over elevated baseline values that were stable or decreasing or development of new pathological Q waves in at least 2 contiguous leads on the electrocardiogram. Symptoms of cardiac ischemia were not required.
Time Frame: Up to 30 plus or minus (+-) 5 days after the catheter ablation procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Number analyzed (Participants) | 114 | 107
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Ischemic Stroke
Description: Stroke was defined as a new, sudden, focal neurological deficit resulting from a presumed cerebrovascular cause that was not reversible within 24 hours and not due to a readily identifiable cause such as a tumor or seizure.
Time Frame: Up to 30 plus or minus (+-) 5 days after the catheter ablation procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Number analyzed (Participants) | 114 | 107
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Non-Central Nervous System (Non-CNS) Systemic Embolism
Description: The Non-CNS systemic embolism was defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms, (example; trauma, atherosclerosis, instrumentation).
Time Frame: Up to 30 plus or minus (+-) 5 days after the catheter ablation procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Number analyzed (Participants) | 114 | 107
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Vascular Death
Description: Any death that was not clearly non-vascular. Examples of vascular death included deaths due to bleeding, Myocardial Infarction (MI), stroke, heart failure and arrhythmias.
Time Frame: Up to 30 plus or minus (+-) 5 days after the catheter ablation procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Number analyzed (Participants) | 114 | 107
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Screening up to Week 8-10
Description: The overall treatment-emergent adverse event (TEAEs), serious adverse events, and adverse events leading to discontinuation are based on 244 participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Rivaroxaban | Vitamin K Antagonist
Serious Adverse Events (participants affected / at risk) | 17/123 | 20/121
Other Adverse Events (participants affected / at risk) | 26/123 | 20/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=123) | Vitamin K Antagonist (N=121)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 5
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Sinus arrest (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Puncture site haemorrhage (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 2
International normalised ratio increased (Investigations) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Atonic seizures (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=123) | Vitamin K Antagonist (N=121)
Atrial fibrillation (Cardiac disorders) | 10 | 10
Fatigue (General disorders) | 8 | 2
Haematoma (Vascular disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.